CLINICAL TRIAL: NCT04230408
Title: Intensified Chemo-immuno-radiotherapy With Durvalumab (MEDI4736) for Stage III Non-Small Cell Lung Cancers (NSCLCs): a Brazilian Single Arm Phase II Study (PACIFIC BRAZIL)
Brief Title: Intensified Chemo-immuno-radiotherapy With Durvalumab for Stage III Non-Small Cell Lung Cancers
Acronym: PACIFIC BRAZIL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: AstraZeneca (Industry); Libbs Farmacêutica LTDA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LACOG 2218
Record Dates: First submitted 2020-01-10; First posted 2020-01-18 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Lung Neoplasms
Keywords: Stage III Non-Small Cell Lung Cancer; Unresectable Non-Small Cell Lung Cancer; Durvalumab; MEDI4736
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Prospective single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DURVALUMAB (MEDI4736) + carboplatin-paclitaxel (Experimental): Induction chemo-immunotherapy phase:
  Two cycles of Paclitaxel 200 mg/m2, Carboplatin AUC 6 and Durvalumab 1500 mg intravenously every 21 days.
  Concurrent chemo-immuno-radiotherapy phase:
  Radiation therapy concomitantly with: paclitaxel 50 mg/m2 intravenously every 7 days (+/- 3 days) until completion of radiation therapy, carboplatin AUC 2 intravenously every 7 days (+/- 3 days) until completion of radiation therapy and durvalumab 1500 mg intravenously every 21 days (+/- 6 days) for a maximum of 2 doses.
  Concurrent chemo-immuno-radiotherapy:
  Durvalumab 1500 mg intravenously every 28 days (+/- 7 days) for a maximum of 12 doses
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Intensified chemo-immuno-radiotherapy with durvalumab in combination with carboplatin, paclitaxel and radiation
  Other Names: Carboplatin; Paclitaxel

SUMMARY:
This is a phase II study that will assess if Durvalumab (MEDI4736) used as induction chemo-immunotherapy followed by concurrent chemo-immuno-radiotherapy and consolidation immunotherapy may improve oncologic outcomes compared with standard of care chemoradiation followed by durvalumab (as in the PACIFIC trial) with a reasonable safety profile.

DETAILED DESCRIPTION:
Prospective, non-randomized, open label, single arm, multi-institutional, phase 2 study, including patients with stage III non-small cell lung cancer able to receive concurrent chemoradiation. Eligible patients will then receive treatment as follows:

Induction chemo-immunotherapy Two 21-day cycles of carboplatin, paclitaxel and durvalumab will be given BEFORE concurrent chemo-immuno-radiotherapy.

Thereafter, patients without progressive disease (or patients with disease progression that is still locally advanced and can be safely encompassed within tolerable radiation fields) will receive concurrent chemo-immuno-radiotherapy, as follows:

Concurrent chemo-immuno-radiotherapy Concurrent carboplatin, paclitaxel, and durvalumab with radiation therapy, initiated preferably 3-5 weeks after the last dose of induction chemo-immunotherapy.

Thereafter, patients without progressive disease will receive consolidation immunotherapy, as follows:

Consolidation immunotherapy Twelve 28-day cycles of durvalumab will be given, initiated preferably within one week following concurrent chemo-immuno-radiotherapy.

ELIGIBILITY:
INCLUSION CRITERIA

1. Histologically or cytologically confirmed non-small cell lung cancer.
2. Stage III according to the American Joint Committee on Cancer (AJCC) Staging Manual, 8th edition.
3. No prior systemic therapy, radiation therapy, or surgery for the current cancer.
4. Age ≥ 18 years at time of study entry
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Body weight >30kg
7. Pre- or post-bronchodilator forced expiratory volume 1 ≥ 1.2 litres/second or ≥ 50% of predicted value
8. Adequate normal organ and marrow function

EXCLUSION CRITERIA

1. Patients whose radiation treatment is likely to encompass a volume of whole lung receiving ≥ 20 Gy in total of more than 35% of lung volume.
2. Patients whose radiation treatment is likely to deliver a cardiac dose V50 > 25%
3. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
4. Participation in another clinical study with an investigational product with anti-neoplastic activity during the last 3 weeks prior to treatment initiation
5. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
6. History of allogenic organ transplantation.
7. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
8. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab.
9. Prior randomisation or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
10. Patients who have received prior anti-PD-1, anti PD-L1 or anti CTLA-4 antibodies
11. Receipt of live attenuated vaccine within 30 days prior to the first dose of investigational product.
12. Prior radiation therapy to the region of the study cancer that would result in overlap of radiation therapy fields.
13. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of the investigational product.
14. Active or prior documented autoimmune or inflammatory disorders
15. Uncontrolled intercurrent illness
16. History of another primary malignancy
17. Known active infection including tuberculosis , hepatitis B, hepatitis C, or human immunodeficiency virus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
12 months Progression-Free Survival | Tumor scans will be performed at baseline, after the induction and concomitant phases and 3, 6, 9, and 12 months after the last dose of radiation therapy.
  Proportion of patients who are alive and progression-free 12 months after cycle 1, day 1 of induction treatment, estimated by the Kaplan-Maier method and using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Overall Survival (OS) | OS will be evaluated until month 24 after C1D1.
  Time from cycle 1, day 1 of induction treatment until death due to any cause.
Overall response rate to induction treatment | Tumor scans will be performed at baseline, after the induction and concomitant phases and 3, 6, 9, and 12 months after the last dose of radiation therapy.
  The proportion of patients with at least one tumor scan of complete response (CR) or partial response (PR) using RECIST v1.1.
Patterns of Failure | Tumor scans will be performed at baseline, after the induction and concomitant phases and 3, 6, 9, and 12 months after the last dose of radiation therapy.
  Rate of disease failure in local, regional and distant sites

CONTACTS AND LOCATIONS:
Locations (6):
- Brazil (6):
  - INCA, Rio de Janeiro, Rio de Janeiro
  - Liga Norte Riograndense Contra o Câncer, Natal, Rio Grande do Norte
  - CPO, Porto Alegre, Rio Grande do Sul
  - COI Américas, Rio de Janeiro
  - Beneficiencia Portuguesa de São Paulo/Hospital São José, São Paulo
  - ICESP, São Paulo